CLINICAL TRIAL: NCT00973752
Title: Treatment of Older Adults With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Beth Israel Deaconess Medical Center (Other); Enzon Pharmaceuticals, Inc. (Industry); Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Amir Fathi, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-356
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Prednisone; Vincristine; Doxorubicin; pegaspargase; Cytarabine; Methotrexate; Imatinib Mesylate; Clofarabine; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental): All patients treated on same arm
  Interventions: Drug: Prednisone; Drug: Vincristine; Drug: Doxorubicin; Drug: PEG-asparaginase; Drug: Cytarabine; Drug: Methotrexate; Drug: Imatinib; Drug: Clofarabine; Drug: 6 Mercaptopurine

INTERVENTIONS:
Drug: Prednisone — Orally during Induction, Consolidation 1, CNS, Consolidation 2, and Continuation therapy.
Drug: Vincristine — Intravenously during Induction, CNS, Consolidation 2 and Continuation Therapy
Drug: Doxorubicin — Intravenously during Induction, CNS, and Consolidation 2 therapy
Drug: PEG-asparaginase — Intravenously during Induction, Consolidation 1, CNS, and Consolidation 2 therapy
Drug: Cytarabine — Intrathecally during Induction and CNS therapy
Drug: Methotrexate — Intrathecally during Induction, CNS, and Continuation Therapy
Drug: Imatinib — Orally during Induction, Consolidation 1, CNS, Consolidation 2 and Continuation Therapy
Drug: Clofarabine — Intravenously during Consolidation 1 Therapy
Drug: 6 Mercaptopurine — Orally during CNS, Consolidation 2 and Continuation Therapy

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of a multi-drug regimen (which includes prednisone, vincristine, cytarabine, doxorubicin, 6 mercaptopurine, and methotrexate) which is considered standard treatment for children and young adults with acute lymphoblastic leukemia (ALL), in combination with PEG-asparaginase and clofarabine to treat older adults with ALL. PEG-asparaginase has been used in chemotherapy treatment regimens for both children and adults with ALL. Clofarabine has been used in chemotherapy treatment regimens for children with ALL and has been shown to decrease the number of leukemia cells. Participants with leukemia that has an abnormal chromosome, called the Philadelphia chromosome, will also be given imatinib.

DETAILED DESCRIPTION:
* This research study has stages of treatment as follows: 1) Induction 2) Consolidation 1 3) Stem cell of Bone Marrow Transplant (if the participant is eligible). If the participant does not have a transplant: 4) CNS Therapy 5) Consolidation 2 6) Continuation Therapy.
* During all phases of study treatment, participants will have additional tests and procedures to monitor their health and for research purposes. These tests will include: physical exams, blood tests, bone marrow aspirate/biopsy and EKGs (electrocardiogram) and/or ECHOs (echo-cardiogram).
* INDUCTION STAGE: This stage lasts for about one month. The study drugs and the way they are administered are as follows: Prednisone orally on days 1-21 for participants less than 60 and days 1-7 for participants 60 or greater; Vincristine intravenously on days 1, 8, 15 and 22; Doxorubicin intravenously on days 1 and 2; PEG-Asparaginase intravenously on days 7 and 21; Cytarabine intrathecally on day 1; Methotrexate intrathecally on day 29; Imatinib orally on days 14-29 if participant has the Philadelphia Chromosome.
* After induction, if there is evidence of ALL in the spinal fluid, participants may need to receive more intrathecal therapy.
* CONSOLIDATION 1 Therapy: This stage will last about one month. Participants will receive Consolidation 1 Therapy, regardless of whether or not their ALL is in full remission after Induction. The study drugs and the way they are administered are as follows: Prednisone orally days 1-5; Clofarabine intravenously days 1-5; PEG-Asparaginase intravenously days 1 and 15; Imatinib continues orally for participants with the Philadelphia Chromosome.
* After the participants blood counts return to normal, their bone marrow will be tested. If the bone marrow shows remission, participants will proceed to the next stage of the study. If the bone marrow does not show remission, the participants will no longer continue on this study.
* STEM CELL or BONE MARROW TRANSPLANTATION: The next stage is stem cell or bone marrow transplantation if the participant is eligible. If the participant receives a stem cell transplant, they will receive additional chemotherapy (separate from the study drugs) followed by an infusion of stem cells. If the participant receives a bone marrow transplant, they will have a bone marrow aspirate and biopsy 3 months after the transplant and 12 months from the start fo the induction to monitor the status of the ALL. If the participant receives a bone marrow or stem cell transplant, they will continue to be a part of the study, but will not proceed with CNS Therapy, Consolidation 2 Therapy, and Continuation Therapy.
* CENTRAL NERVOUS SYSTEM (CNS) THERAPY: CNS therapy will begin between 2 and 6 weeks following the end of Consolidation 1. This stage will last about one month. The study drugs and the way they are administered are as follows: vincristine intravenously on day 1; doxorubicin intravenously on day 1; 6 mercaptopurine orally on days 1-14; prednisone orally on days 1-5; PEG-asparaginase intravenously on days 1 and 15; methotrexate/cytarabine/prednisone intrathecally weekly for 3 weeks; imatinib orally continues daily if the participant has the Philadelphia Chromosome.
* Radiation therapy will also be given during this stage of the participant is under 60 years old. The purpose of radiation therapy is to prevent ALL from coming back in the brain. Radiation will be given in 8 treatments, given once a day, and will be scheduled with other study treatment.
* CONSOLIDATION 2 THERAPY: This stage begins as soon as CNS Therapy ends and lasts about 8 months. Participants will receive repeated cycles of the study drug treatment about every 4 weeks. The study drugs and the way they are administered are as follows: vincristine intravenously on day 1; doxorubicin intravenously on day 1; 6 mercaptopurine orally on days 1-14; prednisone orally days 1-5; PEG-asparaginase orally on days 1 and 15 (first cycle only); imatinib orally continues daily if the participant has Philadelphia chromosome.
* CONTINUATION THERAPY: This stage begins at the end of Consolidation 2 Therapy. The goal of this stage is to get rid of all of the ALL in the body. Participants will receive repeated cycles of the study drug treatment every 4 weeks. It will last until the participant has been in remission for 2 years. The study drugs and the way they are administered are as follows: vincristine intravenously on day 1; mercaptopurine orally on days 1-14; prednisone orally on days 1-5; methotrexate intravenously on day 15; imatinib orally continues daily if the participant has Philadelphia chromosome.

ELIGIBILITY:
Inclusion Criteria:

* Acute lymphoblastic leukemia, excluding known mature B-cell ALL by the presence of any of the following: surface immunoglobulin, L3 morphology, t(8;14)(q24;q32), t(8;22), or t(2;8).
* Patients with mature B-cell ALL will be removed from the protocol as soon as the diagnosis is made and should be treated on a B-cell leukemia protocol.
* Patients with lymphoblastic lymphoma are also eligible
* No prior anti-leukemic therapy except <1 week of steroids, and/or emergent radiation therapy to the mediastinum, or hydroxyurea or emergent leukopheresis. Longer steroid use for diseases other than leukemia is permitted.
* Age 51-75 years
* Ejection fraction > 45%
* Creatinine < 2.0 mg/dl
* Total bilirubin < 3.0 mg/dl
* ECOG (Eastern Cooperative Oncology Group) Performance Status of 0, 1, 2
* Non-pregnant and non lactating

Exclusion Criteria:

* Known HIV positive
* Comorbid medical condition, in the investigator's opinion, would make participation in this trial and adherence to the protocol guidelines difficult
* Active psychiatric or mental illness making informed consent or careful clinical follow-up unlikely

Ages: 51 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-08; Primary Completion 2014-12 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Fathi, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Fathi AT, DeAngelo DJ, Stevenson KE, Kolitz JE, Asch JD, Amrein PC, Attar EC, Steensma DP, Wadleigh M, Foster J, Connolly C, Galinsky I, Devoe CE, Stone RM, Neuberg DS, Ballen KK. Phase 2 study of intensified chemotherapy and allogeneic hematopoietic stem cell transplantation for older patients with acute lymphoblastic leukemia. Cancer. 2016 Aug 1;122(15):2379-88. doi: 10.1002/cncr.30037. Epub 2016 May 12. PMID 27171984

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: All patients treated on same arm
  Prednisone: Orally during Induction, Consolidation 1, CNS (central nervous system), Consolidation 2, and Continuation therapy.
  Vincristine: Intravenously during Induction, CNS, Consolidation 2 and Continuation Therapy
  Doxorubicin: Intravenously during Induction, CNS, and Consolidation 2 therapy
  PEG-asparaginase: Intravenously during Induction, Consolidation 1, CNS, and Consolidation 2 therapy
  Cytarabine: Intrathecally during Induction and CNS therapy
  Methotrexate: Intrathecally during Induction, CNS, and Continuation Therapy
  Imatinib: Orally during Induction, Consolidation 1, CNS, Consolidation 2 and Continuation Therapy
  Clofarabine: Intravenously during Consolidation 1 Therapy
  6 Mercaptopurine: Orally during CNS, Consolidation 2 and Continuation Therapy
Period: Overall Study
Arm/Group | Experimental
Started | 30
Completed | 30
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 58 [51 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 27
  Not Available | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
White blood cell count [Median (Full Range); unit: 10^3 cell per μL] | 10.4 [0.7 to 570]
Performance status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group Performance Status 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any self-care totally confined to bed or chair
  5. Dead
  Participants
    ECOG 0 | 14
    ECOG 1 | 11
    ECOG 2 | 5
Chromosomal alterations [Count of Participants; unit: Participants]
  Philadelphia chromosome positive | 12
  Mixed lineage leukemia rearrangement | 2
Immunophenotype [Count of Participants; unit: Participants] — acute lymphoblastic leukemia (ALL) immunophenotype
  Participants
    B-cell ALL | 29
    T-cell ALL | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at One Year
Description: The number of participants alive one year after baseline.
Time Frame: 1 years
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 30
Participants | 19

ADVERSE EVENTS:
Arm/Group | Experimental
Serious Adverse Events (participants affected / at risk) | 10/30
Other Adverse Events (participants affected / at risk) | 18/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=30)
Infection w/ gr. 3/4 neutropenia (Infections and infestations) | 7
Infection - other (Infections and infestations) | 3
Allergic Reaction (Immune system disorders) | 3
Transaminitis (Hepatobiliary disorders) | 7
Hyperbilirubinemia (Hepatobiliary disorders) | 10
Azotemia (Renal and urinary disorders) | 1
Tumor lysis syndrome (General disorders) | 2
stomatitis (Gastrointestinal disorders) | 1
Gastrointestinal bleeding (Gastrointestinal disorders) | 2
Neuropathy (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental (N=30)
Grade 2 Anemia (Blood and lymphatic system disorders) | 12 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Allergic reaction (Immune system disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Hypertension (Cardiac disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 hypotension (Cardiac disorders) | 6 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 fatigue (General disorders) | 18 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Insomnia (General disorders) | 2 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 weight loss (General disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 erythema multiforme (Skin and subcutaneous tissue disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 pruritis (Skin and subcutaneous tissue disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 rash (Skin and subcutaneous tissue disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 anorexia (Gastrointestinal disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 colitis (Gastrointestinal disorders) | 2 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 constipation (Gastrointestinal disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 diarrhea (Gastrointestinal disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 stomatitis (Gastrointestinal disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 nausea (Gastrointestinal disorders) | 11 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 taste alteration (Gastrointestinal disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 vomiting (Gastrointestinal disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 febrile neutropenia (Infections and infestations) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Infection (Infections and infestations) | 9 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Edema (General disorders) | 9 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 transaminitis (Hepatobiliary disorders) | 7 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Elevated alkaline phosphatase (Hepatobiliary disorders) | 2 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Hyperbilirubinemia (Hepatobiliary disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 azotemia (Renal and urinary disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 hyperglycemia (Metabolism and nutrition disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 hypoalbuminemia (General disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 hypocalcemia (Metabolism and nutrition disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 weakness (General disorders) | 4 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 mental status change (General disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 neuropathy (Nervous system disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 Abdominal pain (Gastrointestinal disorders) | 5 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 back pain (General disorders) | 2 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 pain, other (General disorders) | 3 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol
Grade 2 ureteral obstruction (Renal and urinary disorders) | 1 — Grade 1 toxicities were not required to be reported per protocol

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes